CLINICAL TRIAL: NCT01611025
Title: The Impact on the Hospital's Microbial Ecology Follow the Introduction of Ertapenem and Other Newly Introduced Antibiotic, Using Antibiotic Utilization and Hospital Susceptibility Data Over Time
Brief Title: Hospital Microbial Ecology Follow the Introduction of Ertapenem and Other Newly Introduced Antibiotic Over Time
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: MISP39134
Record Dates: First submitted 2011-10-01; First posted 2012-06-04 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Infectious Diseases
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective, multicentre, observational study to assess the trends in antibiotic utilization and hospital ecology with respect to susceptibility patterns of selected bacterial isolates to the utilized antibiotics.

DETAILED DESCRIPTION:
This is a retrospective, multicentre, observational study to assess the trends in antibiotic utilization and hospital ecology with respect to susceptibility patterns of selected bacterial isolates to the utilized antibiotics.

There will be two sets of data collected: Hospital acquired infection (only the first pathogen cultured of each episode) and All infection (the whole hospital susceptibility data)

Primary Objectives:

1. To study the impact of the introduction of ertapenem on the susceptibility pattern of various pathogens to imipenem/meropenem.
2. To study the impact of the introduction of ertapenem on the susceptibility of all Gram negative bacilli to antimicrobial agents commonly used in the participated study sites.
3. To explore the trend in antimicrobial utilization before and after the introduction of new antimicrobial agents to the hospital formulary during the index period.

Secondary Objectives:

1. To study the trend of antimicrobial susceptibility to ESBL-producing Enterobacteriaceae during the index period
2. To study the impact of the introduction of other newly introduced antibiotics (e.g., tigecycline) on the susceptibility pattern of various pathogens to carbapenems
3. To study the prevalence and trend of Pan drug resistant Acinetobacter baumannii and Pseudomonas aeruginosa resistant during the index period

Exploratory objectives:

1) To explore the resistant rates of ESBL-producing Enterobacteriaceae, Pan drug resistant Acinetobacter baumannii and Pseudomonas aeruginosa in different hospitals after adjusted DDD.

Hypotheses:

1. There will be no increase in the utilization rates of other antibiotics, specifically the other carbapenem drugs (imipenem, meropenem) in the index period (2-3 years before and 2-3 years after the introduction of ertapenem).
2. The introduction of ertapenem to the institution formulary will not negatively impact the susceptibility of selected bacterial isolates to the other carbapenem antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* the susceptibility of Pseudomonas aeruginosa
* the susceptibility of Escherichia coli (ESBL and Non-ESBL producing strains)
* the susceptibility of Klebsiella pneumoniae(ESBL and Non-ESBL producing strains)
* the susceptibility of Enterobacter cloacae
* the susceptibility of Enterobacter aerogenes
* the susceptibility of Acinetobacter baumannii
* antibiotic utilization data of carbapenems: Ertapenem, Meropenem, Imipenem
* antibiotic utilization data of Penicillins: Piperacillin/Tazobactam
* antibiotic utilization data of cephalosporins: Ceftriaxone, Cefotaxime, Flomoxef, Cefoperazone, Ceftazidime, cefepime, Cefpirome
* antibiotic utilization data of Aztreonam,
* antibiotic utilization data of fluoroquinolones: Ciprofloxacin, Levofloxacin
* antibiotic utilization data of aminomethylcyclines: Tigecycline

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: selected bacterial isolates, such as but not limited to Pseudomonas aeruginosa, Acinetobacter Baumannii and Enterobacteriaceae species
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2011-06; Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Der Wang, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan